CLINICAL TRIAL: NCT03884725
Title: Profilatic Fibrinogen Concentrate Reduces Postoperative Bleeding in Pediatric Cardiac Surgery With Cardiopulmonary Bypass: Randomized Study
Brief Title: Fibrinogen Concentrate In Children Cardiac Surgery 2
Acronym: FiCCS2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Filomena R B G Galas (Other Government)
Responsible Party: Sponsor-Investigator, Filomena R B G Galas, Associate Professor of Anesthesiology at University São Paulo Medical School, Instituto do Coracao
Organization: Instituto do Coracao (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3864.12.120
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: C.Surgical Procedure; Cardiac; Blood Coagulation Disorders; Hypofibrinogenemia
Keywords: Cardiac surgical procedures; Fibrinogen; Bleeding
MeSH Terms: conditions — Blood Coagulation Disorders; Afibrinogenemia; Hemorrhage | interventions — Fibrinogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fibrinogen concentrate (Active Comparator): patients randomized to fibrinogen group receive intravenous infusion of drug prepared based on ROTEM measurement of maximum clot firmness (MCF)
  Interventions: Drug: Fibrinogen Concentrate
- control (Placebo Comparator): patients randomized to the control group will receive the infusion of 0.9% saline (SF0,9%) prepared based on ROTEM measurement of maximum clot firmness (MCF)
  Interventions: Other: control

INTERVENTIONS:
Drug: Fibrinogen Concentrate — Fibrinogen Concentrate is to be administered as an intravenous infusion after discontinuation of cardiopulmonary bypass and administration of protamine. Subjects are to be given Fibrinogen Concentrate at an individually determined dose based on FIBTEM MCF and body weight as follows: (15 [mm] - MCF [mm]) * body weight [kg] / 140 [mm*kg/g] = gram fibrinogen to be dosed as Fibrinogen Concentrate. Fibrinogen Concentrate is to be infused over 1 to 2 minutes. After Fibrinogen Concentrate infusion, bleeding treatment will follow the predefined, standardized treatment regimen.
  Arms: fibrinogen concentrate
Other: control — 0.9% saline is to be administered as an intravenous infusion after discontinuation of cardiopulmonary bypass and administration of protamine. Patients randomized to the control group will receive the infusion of 0.9% saline (SF0,9%) prepared based on ROTEM measurement of maximum clot firmness (MCF). 0.9% saline is to be infused over 1 to 2 minutes. After 0.9% saline infusion, bleeding treatment will follow the predefined, standardized treatment regimen.
  Arms: control

SUMMARY:
The purporse of this study is evaluate whether fibrinogen concentrate reduces postoperative bleeding in pediatric cardiac surgery with cardiopulmonary by-pass.

DETAILED DESCRIPTION:
Cardiac surgery in children may be associated with excessive perioperative bleeding. Perioperative excessive bleeding is associated with need of transfusion with allogeneic blood products such as red blood cells, fresh frozen plasma, platelet pools, and cryoprecipitate. Furthermore, bleeding may result in re-exploration, which is associated with increased morbidity and mortality.Recent studies have shown that patients and children undergoing cardiac surgery with pump often experience a significant drop in their levels and function of fibrinogen, and it would be in part responsible for the bleeding. Fibrinogen concentrate (Haemocomplettan P)may reduce perioperative bleeding, requirements of blood transfusion and clinical outcomes in children undergoing cardiac surgery with pump.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery with pump
* Written informed consent
* Age under 28 days of life or RACHS-1 equal or greater than 3 or reoperation with age under 10 years

Exclusion Criteria:

* Coagulopathy (INR > 1.5)
* Low platelet count (lower than 100.000)
* Product or albumin allergy
* Active endocarditis
* Blalock-Taussig
* Heart transplant
* Anemia (hemoglobin < 10 g/dL)
* Impossibility to receive blood transfusion
* Hepatic dysfunction (total bilirubin > 1.5 mg/dL)
* Known or suspected hypersensitivity to fibrinogen concentrate
* Thrombophilia or previous thrombosis
* Participation in another study

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
The amount of postoperative bleeding | Within 7 days after cardiac surgery
  The amount of blood loss (tube drainage) in the first 6 hours of ICU admission and daily until the seventh day of ICU. Re-exploration is mandatory if the patient presente excessive bleeding not responsive to clinical measures (warming, coagulopathy correction and/or thrombocytopenia correction), associated hemodynamic instability or evidence of cardiac tamponade.

SECONDARY OUTCOMES:
The amount and type of blood transfusion | within 7 days after cardiac surgery
  The amount and type of intraoperative blood transfusion within the first 6 hours of ICU admission and daily up to the seventh day of ICU.
Rate of acute kidney injury | within 28 days after cardiac surgery
  According to pediatric RIFLE, will be measured daily.
Rate of cardiac complications | within 28 days after cardiac surgery
  Occurrence of arrhythmias, low cardiac output, cardiogenic shock and the need of postoperative ventricular assistance
Rate of neurological complications | within 28 days after cardiac surgery
  Incidence of stroke
Rate of infection complications | within 28 days after cardiac surgery
  Infection (surgical wound infection, pneumonia, urinary tract infection and bloodstream infection), sepsis, severe sepsis and septic shock.
Correlation between clot firmness (FIBTEM) and plasma fibrinogen | After the cardiopulmonary bypass (CPB) weaning and after drug administration during the surgery.
  Relationship among the results of FIBTEM-A10 and plasma fibrinogen level will be performed at the same time
Evaluation of the clot firmness before and after the intervention | After the cardiopulmonary bypass (CPB) weaning and after drug administration during the surgery.
  Evaluation between FIBTEM-A10 that will be measured after the cardiopulmonary bypass (CPB) weaning and after drug intervention
Evaluation of plasma fibrinogen before and after the intervention | After the cardiopulmonary bypass (CPB) weaning, after drug administration during the surgery and in ICU admission.
  Evaluation between the fibrinogen level that will be measured after the cardiopulmonary bypass (CPB) weaning, after drug intervention and in the ICU admission.
Duration of mechanical ventilation | within 28 days after cardiac surgery
  number of hours in which the patient reiman intubated between the date of surgery and discharge from the ICU
Length of vasoactive drugs | within 28 days after cardiac surgery
  number of hours in which the patient will use vasoactive drugs between the date of surgery and discharge from the ICU
Length of ICU stay | within 28 days after cardiac surgery
  number of days between the admission and discharge from the ICU.
Length of hospital stay | within 28 days after cardiac surgery
  number of days between the date of surgery and hospital discharge.
Rate of mortality | within 28 days after cardiac surgery
  Death from all causes occurring up to 28 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Filomena RG Galas, Principal Investigator — University of Sao Paulo
Locations (1):
- Incor - Heart Institute - University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Result] Galas FR, de Almeida JP, Fukushima JT, Vincent JL, Osawa EA, Zeferino S, Camara L, Guimaraes VA, Jatene MB, Hajjar LA. Hemostatic effects of fibrinogen concentrate compared with cryoprecipitate in children after cardiac surgery: a randomized pilot trial. J Thorac Cardiovasc Surg. 2014 Oct;148(4):1647-55. doi: 10.1016/j.jtcvs.2014.04.029. Epub 2014 Apr 18. PMID 24951020
- See also: Bleeding, Bleeding Disorders, Heart Surgery — https://www.nlm.nih.gov/medlineplus/
- See also: Fibrinogen Concentrate — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp